CLINICAL TRIAL: NCT05712512
Title: Early Identification of Autism Spectrum Disorder: Towards an Integrated Biomarker Approach
Brief Title: Experimental Techniques for Early Identification of Autism
Status: Completed | Type: Observational
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Other Study IDs: 845
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Autism Spectrum Disorder; Infant Development
Keywords: siblings; biomarker; autism; infants
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Infant siblings of children with autism spectrum disorder
  Interventions: Behavioral: Neurodevelopmental assessment; Other: Electrophysiological and eyetracking recordings

INTERVENTIONS:
Behavioral: Neurodevelopmental assessment — individual behavioral and socio-communicative assessment from 6 to 36 months
Other: Electrophysiological and eyetracking recordings — Investigation of neural and behavioral biomarkers of autism from 6 to 24 months

SUMMARY:
This project deals with essential challenges in the context of Autism Spectrum Disorder, benefiting from a longitudinal design in infancy and a cutting-edge electroencephalogram/eye-tracking integrated approach. The investigators will focus on multisensory audiovisual integration to identify early markers of autism in infants at-risk for autism. The investigators will characterize early derailments from the typical developmental trajectories to identify critical "time windows" and better describe the heterogeneity of autism.

DETAILED DESCRIPTION:
Autism Spectrum Disorder is a heterogeneous condition characterized by atypical social communication and repetitive patterns of behavior, with recent Italian prevalence estimates of one in 77. The heterogeneity of autism is expressed in individual variation not only in the severity of core symptoms but also in cognitive, language, and behavioral skills, which show different developmental trajectories. Moreover, there is a strong interest in identifying reliable behavioral and brain-based predictors, which may constitute useful tools for early detection of at-risk cases. In particular, autistic individuals perform poorly during conditions that require integration across multiple sensory modalities such as audiovisual sensory integration, and process differently social and non-social stimuli compared to neurotypical counterparts.

However, the study of potential interaction between sensory and social processing in the first years of life is still scarce. No study examined early social and sensory markers in infant siblings of autistic children using integrated experimental techniques.

The study includes siblings of autistic children and neurotypical toddlers recruited at 18 months and a follow-up evaluation is collected at 24 months. At both time-points, all children are assessed with an experimental protocol, including behavioral and neurophysiological measures.

The integrated electroencephalogram -eyetracking task focuses on sensory processing in social (face saying "wow" in infant-directed speech) and non-social (spinning top toy) conditions. Presented videos are presented both in synchronous and asynchronous modalities (1000 ms delay audio presentation). Electroencephalographic signal is recorded by High-Density 128-channel system and pupil dilations are recorded using a Tobii ProSpectrum 300 Hertz system. In addition, complete information about clinical measures is collected for all children at 18 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged between 6 and 36 months
* Toddlers at elevated likelihood of developing autism because siblings of children with autism

Exclusion Criteria:

* gestational age <36 weeks
* Griffiths general quotient < 70
* presence of major complications in pregnancy and/or delivery likely to affect brain development
* presence of neurological deficits, dysmorphic markers, or other medical conditions

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Longitudinal sample of infant siblings of children with autism
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Cognitive outcome of standardized tests | age 36 months
  standardized scores (i.e., Intelligence quotient scores) of Griffiths scales will be measured and will be correlated with electroencephalographic and eyetracking parameters
Socio-communicative outcome of standardized tests | age 36 months
  standardized scores (Calibrated severity scores) of Autism Diagnostic Observation Schedule - 2 edition (Social Affect, Restricted/Repetitive behaviors) will be measured and will be correlated with electroencephalographic and eyetracking parameters
Sensory outcome of standardized tests | age 36 months
  standardized scores (i.e., z-scores) of sensory profile-2 (sensory seeking, avoiding, sensitivity, registration) will be measured and will be correlated with electroencephalographic and eyetracking parameters
Change of electroencephalografic theta power and looking behavior during development | at 6, 12, 18 and 24 months
  Electroencephalographic theta power, looking behavior (time of fixation in different areas of interest, pupillometry parameters) to synchronous/asynchronous audio-visual stimuli will be measured longitudinally.

CONTACTS AND LOCATIONS:
Locations (1):
- Associazione La Nostra Famiglia - IRCCS Eugenio Medea, Bosisio Parini, LC, Italy

IPD SHARING:
Plan to Share IPD: No